CLINICAL TRIAL: NCT06361381
Title: The Combined Effect of Transcutaneous Electrical Nerve Stimulation and Transcutaneous Auricular Vagus Nerve Stimulation on Pressure and Heat Pain Thresholds in Pain-Free Subjects: A Randomized Cross-Over Trial
Brief Title: The Combined Effect of TENS and TaVNS on Pressure and Heat Pain Thresholds in Pain-Free Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Principal Investigator, Richard Liebano, Associate Professor, University of Hartford
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 24-01-281
Record Dates: First submitted 2024-03-25; First posted 2024-04-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Healthy Volunteers
Keywords: Transcutaneous Electric Nerve Stimulation; Transcutaneous Auricular Vagus Nerve Stimulation; Randomized cross-over trial; Pain Measurement; Pain Threshold
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TaVNS (Experimental): Active TaVNS: frequency of 25 Hz, pulse duration of 200 µs, at a strong but comfortable intensity.
  Interventions: Device: Active Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS); Device: Transcutaneous Electrical Nerve Stimulation
- Placebo TaVNS (Placebo Comparator): Placebo TaVNS: the intensity will be increased to a sensory level and then decreased to 0 mA
  Interventions: Device: Placebo Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS); Device: Transcutaneous Electrical Nerve Stimulation

INTERVENTIONS:
Device: Active Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS) — Both concha will be swabbed with an alcohol wipe before applying a thin layer of conductive gel. An ear clip electrode will be placed in the concha of both ears.
  A frequency of 25 Hz will be applied with a pulse duration of 200 µs. Every 5 minutes, the subject will be asked if the intensity can be increased, decreased or remain the same to maintain the same level of intensity. Participants will also receive active TENS, 100 Hz, 200 µsec on forearm.
  Other Names: TaVNS
  Arms: Active TaVNS
Device: Placebo Transcutaneous Auricular Vagus Nerve Stimulation (TaVNS) — For placebo TaVNS, the intensity will be increased to a sensory level and then decreased to 0 mA. Participants will also receive active TENS, 100 Hz, 200 µsec on forearm.
  Other Names: Placebo TaVNS
  Arms: Placebo TaVNS
Device: Transcutaneous Electrical Nerve Stimulation — TENS will be applied on subject's forearm at a strong but comfortable intensity
  Other Names: TENS

SUMMARY:
Transcutaneous electrical nerve stimulation (TENS) is a non-invasive modality that utilizes electrical currents to modulate pain in populations with acute and chronic pain. TENS has been demonstrated to produce hypoalgesic effects in postoperative pain, fibromyalgia, knee osteoarthritis, and healthy subjects. Transcutaneous auricular vagus nerve stimulation (TaVNS) is a non-invasive modality that modulates the vagus nerve by stimulating its auricular branches. The effects of the combination of TENS and TaVNS on producing an analgesic response have not been studied. Considering that TENS and TaVNS both stimulate similar analgesic pathways but through different means of activation, the investigators can hypothesize that a combination of both methods can produce a more pronounced analgesic response. Therefore, the objective of this study is to assess the hypoalgesic effect of a combination of TENS and TaVNS in pain-free subjects.

The study will be a simple crossover design conducted at the University of Hartford. Subjects will be recruited from the University of Hartford population via oral communication, digital flyers, and posters on campus. Thirty participants will undergo two sessions in a crossover manner with one week in between. During one session, the participants will receive TENS with active TaVNS and the other session will be a placebo procedure (TENS with placebo TaVNS). The order of these sessions will be randomized. Importantly, the pressure pain threshold (PPT) and heat pain threshold (HPT) assessors will be blinded to the treatment category. For active TaVNS, a frequency of 25 Hz will be applied with a pulse duration of 200 µs. For placebo TaVNS, the intensity will be increased to a sensory level and then decreased to 0 mA. High frequency TENS of 100Hz will be applied in both sessions, with a pulse duration of 200 µsec, asymmetrical biphasic square waveform, and intensity of maximal tolerance without pain. TENS and TaVNS will be turned on for 30 minutes after a baseline measurement of outcomes. TENS and TaVNS will then be turned off, but the electrodes will remain on until completion of post-treatment assessment. Pressure pain threshold, heat pain threshold, blood pressure, oxygen saturation and heart rate will be tested 4 times: Once pre-intervention, once during intervention, once immediately after the intervention and once 15 minutes post-intervention.

DETAILED DESCRIPTION:
The study will be a simple crossover design with the following two treatments: (1) active TaVNS and (2) placebo TaVNS. Each subject will receive both interventions in random order.

Pressure and Heat pain thresholds will be recorded at baseline, 15 min, 30 min, and 45 min.

ELIGIBILITY:
Inclusion Criteria:

* Absence of pain
* Age 18-40
* Men and women

Exclusion Criteria:

* Neurological diseases
* Severe cardiorespiratory disease
* Pregnancy
* Skin infection or lesions or change in sensation at the TENS or TaVNS application site
* Cancer
* Cardiac pacemaker
* Allergy to electrodes
* Chronic illness or pain
* Use of drugs that affect pain or vagal tone in the past 48 hours prior to data collection

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | 2 weeks
  A digital pressure algometer will measure the pain threshold to deep mechanical stimuli in kPa

SECONDARY OUTCOMES:
Heat Pain Threshold | 2 weeks
  Superficial heat pain sensitivity, in degree Celsius, will be assessed using a handheld thermode.
Heart rate | 2 weeks
  Heart rate (beats per minute) will be assessed using a fingertip pulse oximeter
Oxygen saturation | 2 weeks
  Oxygen saturation in percentage will be assessed using a fingertip pulse oximeter
Blood pressure | 2 weeks
  Systolic and Diastolic Blood pressure in millimeters of mercury will be assessed using a upper arm cuff, blood pressure monitor

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Liebano, PhD, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liebano RE, Awad N, Bellino C, Bray K, Rosentrater H, Roy J, Tate C. The combined effect of transcutaneous electrical nerve stimulation and transcutaneous auricular vagus nerve stimulation on pressure and heat pain thresholds in pain-free subjects: a randomized cross-over trial. Trials. 2024 Jul 31;25(1):516. doi: 10.1186/s13063-024-08352-x. PMID 39085951